CLINICAL TRIAL: NCT01977053
Title: Impact of a Telephonic Monitoring During Neo Adjuvant or Adjuvant Chemotherapy
Brief Title: Impact of a Telephonic Monitoring During Inter-treatment Intervals on Emotional State, Quality of Life and Toxicities, on Neo Adjuvant or Adjuvant Chemotherapy-treated Patients
Acronym: EMOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012/04; 2013-A00506-39 (Other: ID-RCB number)
Record Dates: First submitted 2013-10-22; First posted 2013-11-06 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Non-metastatic Patients With Breast Cancer; Non-metastatic Patients With Colon Cancer; Non-metastatic Patients With Rectal Cancer; Patients Undergoing Adjuvant Chemotherapy
Keywords: breast cancer; colon cancer; rectal cancer; adjuvant chemotherapy; phone calls; emotional states; quality of life
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Standard medical care (No Intervention): Arm A: standard supervision and medical care during an adjuvant chemotherapy treatment in France
- B: telephonic monitoring (Experimental): Arm B: telephonic monitoring during inter-treatment intervals + personalized medical care.
  Interventions: Other: Clinical and psychosocial phone calls

INTERVENTIONS:
Other: Clinical and psychosocial phone calls — The standard medical supervision is defined as follows:
  * Prescription of prophylactics medication (corticoid, antiemetic, cream, mouthwash, etc) at each cycle of chemotherapy.
  * Nominative notebook containing details of chemotherapy administered and medical contacts.
  * Consultations with psycho-oncologist or psychiatrist (if necessary).
  The intervention further comprises: nurse phone calls the 3rd and the 8th day of the first three cycles of treatment, and personalized medical care according to toxicities reported.
  Other Names: medical care including social and psychological domains
  Arms: B: telephonic monitoring

SUMMARY:
In health care, the phone has emerged as a clinical tool in its own right, especially for the development of psychological support to patients and that, in many pathologies. Its potential in the development of psycho-social support was quickly identified.

However, to our knowledge, no prospective, randomized studies have evaluated the impact of a telephone call to both the anxiety and the management of side effects of neoadjuvant or adjuvant chemotherapy.

The patient incomplete care by the hospital system and the general practitioner during chemotherapy, as well as the lack of information and poor preparation and / or management of side effects, are a source of distress and lead to a decrease quality of life for the patient and his family.

We propose to determine on a population of 280 patients, the impact of two phone calls during 3 first inter-treatment intervals on the overall measure of mood states of the patient and his principal caregiver (anxiety, depression, confusion, angry, fatigue, force and interpersonal relation). We will also study the gain in quality of life, on anxiety level, frequency and severity of toxicities, as well as emotional comfort of the procedure.

DETAILED DESCRIPTION:
Cancer is widely associated with the concept of psychological distress in a population of patients subject to numerous stressful events. Between 10 to 50% of patients with cancer and their families suffer from clinically significant psychological disorders.

The existence of a broad continuum of manifestations of distress makes it difficult for clinical evaluation. Underestimated and misjudged, it is not always taken into account appropriately. However, these problems have a direct impact not only on the quality of life of patients but also on their ability to share decisions , adhere to treatment, and therefore to get the best care available for the treatment of their cancer.

Interactions between the presence of psychopathological disorders, quality of life and treatment toxicities will be the focus of this study assessing the impact of telephonic monitoring (targeting clinical, psychological and social objectives) in patients with current chemotherapy.

There are communication difficulties on the distress between the patient and the doctor, in part due to the gap between the perceptions of the patient and the caregiver. Indeed, many studies have highlighted the important differences existing between subjective psychosocial needs of the patient and the physician's ability to detect them. In particular, the study of Fallowfield on nearly 2300 medical consultations shows that only 29% of patients whose threshold of distress is clinically significant are identified by their doctors. Similarly, the synthesis carried out in 2005 by Thorne et al. reported the impact of failures of communication between clinicians and patients on the psychosocial experience of illness and treatment, symptom management, decision making and quality of life.

Justification and research hypothesis

In health care, the phone has emerged as a clinical tool in its own right, especially for the development of psychological support to patients and that, in many pathologies. Its potential in the development of psycho-social support was quickly identified.

However, to our knowledge, no prospective, randomized studies have evaluated the impact of a telephone call to both the anxiety and the management of side effects of neoadjuvant or adjuvant chemotherapy.

The patient incomplete care by the hospital system and the general practitioner during chemotherapy, as well as the lack of information and poor preparation and / or management of side effects, are a source of distress and lead to a decrease quality of life for the patient and his family.

We propose to determine on a population of 280 patients, the impact of two phone calls during the first 3 inter-treatment intervals, the overall measure of mood states (anxiety, depression , confusion , anger , fatigue , vigor and interpersonal ) of the patient and his entourage . We also study the gain in quality of life, anxiety level, frequency and severity of toxicities, as well as emotional comfort of the procedure.

We propose to determine on a population of 280 patients, the impact of two phone calls during the 3 first inter-treatment intervals on the overall measure of mood states of the patient and his principal caregiver (anxiety, depression, confusion, angry, fatigue, force and interpersonal relation). We will also study the gain in quality of life, on anxiety level, frequency and severity of toxicities, as well as emotional comfort of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18.
* Patient surgically-treated or no for non inflammatory breast cancer or for colon cancer or rectal cancer.
* Patient to be treated by neo-adjuvant or adjuvant chemotherapy by 5-fluorouracil, epirubicin and cyclophosphamide (FEC)-docetaxel, docetaxel-cyclophosphamide, 5-fluorouracil/leucovorin with oxaliplatin(FOLFOX) or XELOX. A treatment with trastuzumab is allowed in association.
* Patient never treated by chemotherapy.
* Patient with Performance Status under or equal to 2.
* Patient with adequate hematopoietic, hepatic and cardiac functions according to the investigator.
* Patient having read with the information note and having signed the informed consent.
* Patient beneficiating from French health insurance cover.

Exclusion Criteria:

* Patient with psychological state, geographical remote or social problems that contraindicated the participation into the study according to the investigator.
* Patient that must be treated for a metastatic disease.
* Patient not able to attend all study visits.
* Patient not understanding French.
* Patient who don't have a phone.
* Vulnerable patient: pregnant or breast-feeding women, person deprived of freedom by an administrative or judicial decision, person older than 18 being the object of a legal protection measure or outside state to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2013-09; Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
emotional state (anxiety, depression, confusion, angry, fatigue, force and interpersonal relation) | Change from baseline in POMS-f score at 6 weeks
  comparison of the 2 types of monitoring in terms of overall measure of emotional state (anxiety, depression, confusion, angry, fatigue, force and interpersonal relation) of patients, with Profile of Mood States (POMS-f) questionnaire.

SECONDARY OUTCOMES:
Evolution of emotional states scores | Change from baseline in POMS-f score at 6 weeks; Change from baseline in POMS-f score at 9 weeks and Change from baseline in POMS-f score at 12 weeks
  To compare 2 types of supervision in terms of:
  The difference between the overall scores on the POMS-f before the start of treatment, at each treatment and after 3 courses of treatment
toxicities | up to 15 weeks
  To compare 2 types of supervision in terms of proportion of patients with toxicity during treatment, and the maximum grade observed per patient
quality of life | Change from baseline in EORTC QLQ-C30 score at 6 weeks and Change from baseline in EORTC QLQ-C30 score at 12 weeks
  To compare 2 types of supervision in terms of:
  The quality of life of the patient by the European Organization for Research and Treatment of Cancer Qulity of life questionnaire (EORTC QLQ-C30), before the start of treatment, during the 2nd cycle of chemotherapy and after three courses of treatment
anxiety | up to 15 weeks
  To compare 2 types of supervision in terms of:
  The level of anxiety assessed by the number of visits to psychologists, psychiatrists, the sub-score "Anxiety" obtained in the Hospital Anxiety and Depression State (HADS) questionnaire, the anxiolytics and antidepressants intakes
caregiver mood states | Change from baseline in POMS-f score at 6 weeks; Change from baseline in POMS-f score at 9 weeks and Change from baseline in POMS-f score at 12 weeks
  To compare 2 types of supervision in terms of:
  - The overall scores obtained by the caregiver on the POMS-f before, during and after 3 courses of treatment
patient satisfaction | up to 12 weeks
  To compare 2 types of supervision in terms of overall satisfaction scores obtained by the patient after 3 courses of treatment
relationship between psychosocial criteria and anxiety | up to 15 weeks
  To compare 2 types of supervision in terms of:
  - The relationship between the presence of psychosocial frailty criteria and the level of anxiety for patients in group B (number of visits to psychologists, psychiatrists; anxiolytics and antidepressants intake; HADS anxiety scores)

OTHER OUTCOMES:
intervention cost | up to 15 weeks
  To compare 2 types of supervision in terms of cost of the procedure (cost of consultations with psychologists, psychiatrists, cost of telephone calls)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe FOLLANA, Dr., Principal Investigator — Centre Antoine Lacassagne
Locations (2):
- France (2):
  - Centre Antoine Lacassagne, Nice, Cedex 2
  - Polyclinique St Jean, Cagnes-sur-Mer

REFERENCES:
- [Background] Ganz PA, Kwan L, Stanton AL, Krupnick JL, Rowland JH, Meyerowitz BE, Bower JE, Belin TR. Quality of life at the end of primary treatment of breast cancer: first results from the moving beyond cancer randomized trial. J Natl Cancer Inst. 2004 Mar 3;96(5):376-87. doi: 10.1093/jnci/djh060. PMID 14996859
- [Background] Stanton AL. Psychosocial concerns and interventions for cancer survivors. J Clin Oncol. 2006 Nov 10;24(32):5132-7. doi: 10.1200/JCO.2006.06.8775. PMID 17093275
- [Background] Carlson LE, Bultz BD. Cancer distress screening. Needs, models, and methods. J Psychosom Res. 2003 Nov;55(5):403-9. doi: 10.1016/s0022-3999(03)00514-2. PMID 14581094
- [Background] Pitceathly C, Maguire P. The psychological impact of cancer on patients' partners and other key relatives: a review. Eur J Cancer. 2003 Jul;39(11):1517-24. doi: 10.1016/s0959-8049(03)00309-5. PMID 12855257
- [Background] Vitek L, Rosenzweig MQ, Stollings S. Distress in patients with cancer: definition, assessment, and suggested interventions. Clin J Oncol Nurs. 2007 Jun;11(3):413-8. doi: 10.1188/07.CJON.413-418. PMID 17623625